CLINICAL TRIAL: NCT05338710
Title: Support Via Technology: Living and Learning With Advancing FTD
Acronym: STELLA-FTD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: The Association for Frontotemporal Degeneration (Unknown)
Responsible Party: Principal Investigator, Allison Lindauer, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00022721
Record Dates: First submitted 2022-03-04; First posted 2022-04-21 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Caregivers Burnout; Frontotemporal Dementia
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Intervention Model Description: 8-week single group intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STELLA-FTD study (Experimental): One group only
  Interventions: Other: STELLA-FTD

INTERVENTIONS:
Other: STELLA-FTD — Behavioral intervention for caregivers for those with FTD

SUMMARY:
Much effort over the last several decades has been devoted to developing and implementing psychoeducational interventions for family caregiving partners for those with Alzheimer's and relatedm dementias (ADRD). However, few interventions address the specific needs of care partners for those with frontotemporal degeneration (FTD).

This study tests an intervention to support family caregivers for those with FTD.

DETAILED DESCRIPTION:
Much effort over the last several decades has been devoted to developing and implementing psychoeducational interventions for family caregiving partners for those with Alzheimer's and related dementias (ADRD). However, few interventions address the specific needs of care partners for those with frontotemporal degeneration (FTD), the most common form of dementia in adults under age 60.

Caring for a family member with FTD can affect the psychological, social, and relational health of families. Care partners for those with the disease have higher levels of burden and depression, as well as more sleep disturbances and worse financial strain than care partners for those with ADRD. Psychoeducational interventions can alleviate some of the psychological symptoms associated with dementia caregiving, but few programs have been designed for care partners for persons with FTD. Further, many of the existing programs are inaccessible for families due to distance and cost. The STELLA (Support via TEchnology: Living and Learning with Advancing dementia) intervention is designed to teach ADRD care partners strategies for managing behavioral symptoms associated with dementia. STELLA uses videoconferencing to connect care partners, in their own homes, with experienced Guides (e.g., nurses). The Guides use cognitive behavioral techniques to assist care partners in identifying and implementing strategies to reduce distressing behavioral symptoms in the person with dementia.

Our pilot work found that early versions of STELLA reduced the frequency of behavioral symptoms and care partner reactivity to them. In this study, the investigators will adapt STELLA to specifically address the needs of family care partners for persons with frontotemporal degeneration. Aim 1. Adapt STELLA to the needs of care partners for those with FTD

1. Gather FTD care partner feedback on STELLA and suggestions for tailoring STELLA for FTD
2. Adapt STELLA for FTD care partners based on end-user feedback Aim 2. Assess the feasibility, acceptability and STELLA-FTD with FTD care partners Aim 3. Assess the preliminary efficacy of STELLA-FTD on the primary outcomes: reducing the frequency of behavioral symptoms and care partner reactivity to the symptoms as measured on the Revised Memory and Behavior Problems Checklist (RMBPC).

ELIGIBILITY:
Inclusion Criteria:

* Care Partner for family member, close friend or kin with FTD, primary progressive aphasia, progressive supranuclear palsy or other frontotemporal degenerative dementia
* Must speak English
* Must be able to see and hear the videoconference-based interactions.

Exclusion Criteria:

- Family member does not care for someone with FTD conditions.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lindauer, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Layton Aging and Alzheimer's Disease Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Video-recordings and other data from this study may be shared with other investigators for future research studies. A study ID number will be assigned to each participant. Only the investigators and people involved in the conduct of the study will be authorized to link the ID number to the participants. Other investigators who may receive samples of data for research will be given only the ID number which will not identify participants. However, the video-recordings will show participants' faces. Names and any information discussed during the sessions and focus group will be heard in the audio. The faces, names and audio of any other people who enter the camera zone will also be recorded. The information given for this study will be identifiable and will not be private. Participants receive this information on the information sheet.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data is currently available and will be available indefinitely.
Access Criteria: Data is entered in to access-controlled local repository (#6845) and NACC National Repository.
URL: https://naccdata.org/requesting-data/nacc-data

REFERENCES:
- [Result] Lindauer A, Smith S, Gothard S, Mattek N, Tran L, Mooney A. 'There's no straight line...' a consumer-informed intervention for FTD family care partners: the STELLA-FTD pilot study. Aging Ment Health. 2023 Sep-Oct;27(10):2000-2010. doi: 10.1080/13607863.2023.2250741. Epub 2023 Sep 1. PMID 37655616

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We were able to recruit 16 participants
Groups:
- Intervention Group: There is one intervention group that received the STELLA-FTD intervention. The behavioral intervention was provided to participants and outcomes were measured prior to and after the intervention within the same group.
Period: Overall Study
Arm/Group | Intervention Group
Started | 16
Completed | 13
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: This group received the STELLA-FTD intervention.
Arm/Group | Intervention Group
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16
Rural Status [Count of Participants; unit: Participants]
  Metropolitan | 14
  Rural | 2
Diagnosis of Care Recipient [Count of Participants; unit: Participants] — Dementia diagnosis of care recipients. BvFTD = Behavioral variant FTD; PPA = Primary progressive aphasia; PSP = Progressive supranuclear palsy.
  Participants
    Bv-FTD | 7
    PPA | 7
    PSP | 1
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Revised Memory and Behavior Problems Checklist (RMBPC)
Description: The primary outcome variable, reactivity, will be assessed with the RMBPC, which measures the frequency of care recipient behavioral symptoms and care partner reactions to these behaviors. The RMBPC was chosen because it aligns with our theoretical foundation that assumes burden is a result of care partner reactions to behavioral symptoms.
  The RMBPC is a 29-item caregiver report measure, 5-point Likert scale with frequency measuring from 0 (never occurred) to 4 (daily or more often) and reactivity measuring from 0 (not at all) to 4 (extremely) for a total score between 0-116 for each subscale (frequency subscale and reactivity subscale). Higher scores indicate greater behavioral problems.
Time Frame: Pre-intervention (at Week 1) and Post-Intervention (at Week 8)
Population: thirteen individuals completed this prior to intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Group: RMBPC prior to STELLA-FTD
Arm/Group | Intervention Group
Number analyzed (Participants) | 13
units on a scale
  Pre intervention, behavior frequency | 28.5 (15.9)
  Post intervention; behavior frequency | 25.2 (15.3)
  Pre-intervention, reactivity | 16.6 (12.9)
  Post intervention, reactivity | 15.8 (13.5)

2. Secondary Outcome: Quality of Life Alzheimer's Disease, Care Partner
Description: This is a brief, 13-item measure designed specifically to obtain a rating of the caregiver's Quality of Life. The measure focuses on quality of life domains. It uses simple and straightforward language and responses & includes assessments of the individual's relationships with friends and family, concerns about finances, physical condition, mood, and an overall assessment of life quality. The total range is 13 to 52 with lower scores indicating worse quality of life.
Time Frame: Pre-intervention (at Week 1) and Post-Intervention (at Week 8)
Population: Higher scores= better QoL
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Group: The intervention group that completed STELLA-FTD intervention.
Arm/Group | Intervention Group
Number analyzed (Participants) | 13
units on a scale
  QoL, care partners pre | 37.6 (5.06)
  QoL, care partners, post | 36.2 (3.95)

3. Secondary Outcome: Family Caregiver Self-Efficacy Scale
Description: Measures caregiver self-efficacy for symptoms management and community support service use. Scale 10-100, higher scores indicating better sense of self-efficacy.
Time Frame: Pre-intervention (at Week 1) and Post-Intervention (at Week 8)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Group: Self-efficacy pre-intervention
Arm/Group | Intervention Group
Number analyzed (Participants) | 13
units on a scale
  Self-efficacy pre | 61.1 (18.8)
  Self-efficacy post | 62.8 (18.3)

4. Secondary Outcome: Center for Epidemiologic Studies Depression
Description: This is a 10-item scale that measures depression; the range is 0 (no depression) to 30 (severe depression).
Time Frame: Pre-intervention (at Week 1) and Post-Intervention (at Week 8)
Population: Depression assessed prior to and after study
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Group: Post-intervention, R: This group received the STELLA-FTD intervention
Arm/Group | Intervention Group
Number analyzed (Participants) | 13
units on a scale
  CESD pre | 10.8 (5.78)
  CESD post | 11.3 (6.33)

5. Secondary Outcome: Marwit Meuser Caregiver Grief Index
Description: Caregiver grief; Scale 18-90, higher scores=worse grief
Time Frame: Pre-intervention (at Week 1) and Post-Intervention (at Week 8)
Population: higher scores=higher grief
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Group: received STELLA-FTD
Arm/Group | Intervention Group
Number analyzed (Participants) | 13
units on a scale
  MMCGI pre | 54.2 (13.7)
  MMCGI post | 55.3 (13.7)

6. Secondary Outcome: Caregiver Guilt Questionnaire (CGQ)
Description: The CGQ is a 22-item caregiver report measure, 5-point Likert scale designed to measure guilt in caregivers with response options from 0 (never) to 4 (always or almost always). Items are organized into five main subscales that are scored by computing the sum of the scores of the items belonging to the corresponding scale.
  "Guilt about doing wrong by the care recipient" includes 7 items with a score range of 0-28. "Guilt about failing to meet the challenges of caregiving" includes 6 items with item #6 being reverse scored. The score ranges from 0-24. "Guilt about self-care" includes 4 items with a score range of 0-16. "Guilt about neglecting other relatives" includes 2 items with a score range of 0-8. "Guilt about having negative feelings towards other people" includes 3 items with a score range of 0-12.
  The total score on the CGQ consists of the sum of the scores of all the subscales, with a total score ranging from 0-88. A higher total score reflects greater guilt.
Time Frame: Pre-intervention (at Week 1) and Post-Intervention (at Week 8)
Population: higher scores=greater guilt
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 13
units on a scale
  Negative feelings towards others pre | 2.23 (1.92)
  Negative feelings post | 1.92 (2.43)
  Neglecting other relatives, pre | 2.31 (2.02)
  Neglecting others post | 2.46 (2.63)
  self care efficacy pre | 4.38 (3.8)
  Self care efficacy post | 4.77 (4.21)
  failing to meet challenges pre | 6 (4.6)
  Failing post | 5.85 (4.88)
  Doing wrong by care recipient pre | 9.46 (5.72)
  Doing wrong post | 10.4 (6.24)

7. Secondary Outcome: Experience Survey
Description: Caregiver assessment of program
Time Frame: Post-Intervention (at Week 8)
Population: Count of items
Measure: Number; unit: participants
Groups:
- Intervention Group: Experience survey
Arm/Group | Intervention Group
Number analyzed (Participants) | 13
participants
  It was easy for me to attend | 13
  I could find a safe activity for my family member | 13
  It was easy to connect via Webex | 12
  I had good tech support | 13
  Overall, I was satisfied with the STELLA-FTD experience | 13
  I feel confident that I can use STELLA-FTD skills to manage upsetting behaviors | 13
  I could talk openly with the professionals | 13
  I liked working with other care partners | 13
  I discuss sensitive topics with other care partners | 11

8. Secondary Outcome: Ten-Item Personality Inventory (TIPI)
Description: The Ten-Item Personality Inventory (TIPI) is a 10-item self-report measure of five personality domains: Extraversion, Agreeableness, Conscientiousness, Emotional Stability, and Openness to Experiences. Each item is rated on a 7-point Likert scale ranging from 1 ("Disagree strongly") to 7 ("Agree strongly"). Items 2, 4, 6, 8, and 10 are reverse-scored.
  For this study, items were summed to create a total personality score. Possible total scores range from 10 to 70, with higher scores indicating stronger endorsement of personality characteristics across the five domains (i.e., higher trait expression).
Time Frame: Pre-Intervention (at Week 1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 13
units on a scale | 51 (8.73)

9. Secondary Outcome: Sleep Hygiene Index
Description: The Sleep Hygiene Index (SHI) is a self-administered questionnaire used to assess an individual's sleep hygiene practices. It's a tool used in research and clinical settings to evaluate sleep habits and identify potential areas for improvement. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (always). Total scores range from 0 to 52, with a higher score representing poorer sleep hygiene.
Time Frame: Post-Intervention (at Week 8)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 13
units on a scale | 10.2 (8.66)

10. Secondary Outcome: Contact Survey
Description: A 9-item measure to assess whether caregivers contacted other caregivers or not.
Time Frame: Post-Intervention (at Week 8)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 13
Participants
  Number who did not contact other caregivers | 11
  Number who contacted others | 2

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
The small sample size limited our ability to identify the effect of study intervention on burden in this important caregiving cohort. Limits to classic in-person recruitment strategies due to COVID-19 restrictions made personalized recruitment efforts challenging. This was offset by a multimodal online recruitment strategy that targeted care partners across the western United States.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT05338710/Prot_SAP_001.pdf